CLINICAL TRIAL: NCT04187911
Title: Relationships in Good Hands Trial: Clinical and Cost-effectiveness of Dyadic Developmental Psychotherapy for Abused and Neglected Young Children With Maltreatment-associated Problems and Their Parents
Brief Title: Relationships in Good Hands - Clinical and Cost-effectiveness of Dyadic Developmental Psychotherapy
Acronym: RIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Oxford (Other); University of Nottingham (Other)
Responsible Party: Principal Investigator, Helen Minnis, Professor of Child and Adolescent Psychiatry, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIHR127801; L19083 (Other: NHS R&D Lanarkshire)
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Mental Health; Psychiatric Problems; Child Neglect; Maltreatment; Adoption; Child Behaviour Problem; DDP
Keywords: Feasibility; Randomised; Optimisation; Partnerships; Cost effectiveness; Clinical effectiveness
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Phase 2 Months 10-26 (17 months) To examine the research questions, and minimise bias, we propose to use a single-blind randomised controlled design, with two-groups. The aim of this phase will be to respond to what recruitment and retention rates are over 6 months and trial assessments and intervention acceptability. We will aim to recruit around 60 families.
  Consenting families will be individually randomised 1:1 to DDP or SAU, stratified by site. Individuals who consent to take part will have an equal chance of being randomised to either group.
  Phase 3 (27 months RCT) The third phase will continue as a single-blind individually randomised control superiority definitive trial and will examine clinical and cost-effectiveness of DDP for improving child mental health, compared to SAU. We will aim to recruit additional 180 families. All the procedures will be same as during Phase 2 as explained in details above.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Dyadic Developmental Psychotherapy (DDP) (Experimental): DDP involves approximately twenty 1 hour sessions (usually over 6-9 months) with the adoptive parent/foster carer and child, facilitated by a specifically trained therapist. DDP aims to treat trauma-related problems and Attachment Disorders over about 20 1-hour sessions using the core communication techniques of Playfulness, Acceptance, Curiosity and Empathy (PACE)
  Interventions: Behavioral: Dyadic Developmental Psychotherapy (DDP)
- Control - Services as Usual (SAU) (Active Comparator): SAU tends to be case-dependent with therapists and social workers attempting to respond to the sometimes changeable needs of the family as needs arise.
  Interventions: Behavioral: Services as Usual (SAU)

INTERVENTIONS:
Behavioral: Dyadic Developmental Psychotherapy (DDP) — DDP involves approximately twenty 1 hour sessions (usually over 6-9 months) with the adoptive parent/foster carer and child, facilitated by a specifically trained therapist. The role of the therapist during sessions is to maintain an attuned relationship with both child and parent - modelling and encouraging development of a similarly attuned relationship between the child and parent. Therapists are trained to use Playfulness, Acceptance, Curiosity and Empathy (PACE). Our research suggests that key mechanisms of action in DDP might include the active participation of the parents and increased carer empathy and emotional warmth for the child. DDP experts believe this helps build parental capacity for attuned dialogue with the child, co-creation of the meanings underlying child behaviour, and co-regulation of experienced emotions aiming to address four main problem areas: 1. child emotional regulation 2. parental stress 3. the parent-child relationship 4. child mental health.
  Arms: Intervention - Dyadic Developmental Psychotherapy (DDP)
Behavioral: Services as Usual (SAU) — SAU tends to be case-dependent with therapists and social workers attempting to respond to the sometimes changeable needs of the family as needs arise. At the time of our UK mapping and modelling work, these services were usually CAMHS based. This may have changed, at least for adoptive families, with the advent of the Adoption Support Fund, which, since May 2015, has allowed local authorities / adoption agencies to apply for funding for "essential therapeutic services". A wide range of interventions, many with a scant evidence base, have been purchased - sometimes from private practitioners - since 2015. In addition, relevant NICE guidelines, particularly those on Looked After and Accommodated Children, Attachment and Child Abuse and Neglect, have been published or updated.Our detailed qualitative and quantitative process evaluation throughout all study Phases will be crucial to carefully characterise SAU in all study sites.
  Arms: Control - Services as Usual (SAU)

SUMMARY:
The research question is: Can the research recommend better ways for social care and health services to work work together to help adoptive and foster families? Can a therapy called DDP improve the mental health of 5-12 year old fostered or adopted children? Is DDP worth the commitment families need to give to it - and the extra cost to the services that deliver it? More than half of adopted or fostered children in the UK have mental health problems including ADHD (i.e. hyperactivity, impulsive behaviour and poor concentration), antisocial behaviour and problems with relationships. Abused and neglected children are more likely than others to have problems in school, become homeless, get involved in crime and even die young (e.g. from suicide), yet there are no fully tested treatments for such complex mental health problems. This is a huge problem because early treatment could greatly improve children's life chances - and reduce strain on health and social care budgets.

There is a Dyadic Developmental Psychotherapy (DDP) a parent-child therapy that takes around 20 sessions and focusses on "Playfulness, Acceptance, Curiosity and Empathy". There is not yet available really good evidence for or against it: many UK therapists like DDP, but it is a big commitment for families: once a week for about six months children will need time off school, the parents will need time off work - and this can be hard to explain to school friends, colleagues and bosses. Research team doesn't just need to know if DDP improves children's mental health - they also need to know if the commitment needed is worth it for families and whether the costs to services outweigh the benefits.

In PHASE 1 the research team will find out whether DDP can work smoothly in the three different settings where it is usually delivered: the NHS, Social Care and Private Practice. Many abused children need other medical and psychiatric support so, the research will assess whether children can get any additional assessments or referrals they may need .

In PHASE 2, the research team plans to find out if it is practically possible to run a high quality trial of DDP. This phase will involve 60 families to find out if they are happy to take part (whether offered DDP or usual services). If all goes to plan, these 60 families will contribute to the final results, along with the 180 families involved in the next PHASE 3 when the research team will test whether DDP is better than usual services and, if it is, whether the improvements in child mental health outweigh the costs.

What impact will the research have? This study will make recommendations about how services should work together to help abused and neglected children and their families. If the researcher team finds that DDP is worth the time and money, it could improve the mental health of abused and neglected children across the world.

DETAILED DESCRIPTION:
Abused and neglected children are at extremely high lifetime risk of psychiatric disorder placing a huge burden on health/social care services and society. Virtually all 92,000 children adopted or fostered in the UK have suffered abuse or neglect, therefore risking profoundly negative outcomes in important areas of development including problematic social relationships, academic underachievement and involvement in crime. These disadvantages can lead to negative spirals of poor health and social inequality. Early intervention can greatly improve their life chances, yet there are no adequate psychosocial treatment strategies or care pathways to address the needs of maltreated children. Psychiatric problems of maltreated children are characterised by complexity. They have experienced extreme environmental risk and are at higher genetic risk than peers. Many also struggle to develop and maintain healthy family relationships. Neurodevelopmental disorders such as Attention Deficit/Hyperactivity Disorder (ADHD) and Autism often co-exist with disorders arising from the abuse and neglect such as Conduct Disorder, Attachment Disorders and Post Traumatic Stress Disorder (PTSD) with devastating consequences for lifelong mental health and development. To reflect this complexity, research team uses the overarching term Maltreatment-Associated Psychiatric Problems (MAPP).

The proposed project is a three-phase development and exploratory trial of Clinical and cost-effectiveness of Dyadic Developmental Psychotherapy (DDP) for abused and neglected children with MAPP and their parents compared to Service as Usual (SAU). The data will be collected in 3 phase trial, through a mixture of qualitative and quantitative methods.

Phase 1 Months 1-9 (9 months)

The first phase will focus on intervention and context optimisation that will take place in 3 sites, each representing one of the UK DDP service delivery contexts: NHS, Social Services and Private Practice. The research questions will be addressed through 24-36 qualitative interviews, and focus groups as well as review meetings at each site, with practitioners and managers involved in delivery of DDP and SAU. The research team will require input from the services practitioners and managers but also Young Peoples' Advisory Groups (YPAG) and Patient, Public, Commissioner Involvement (PPCI) groups.

Phase 2 Months 10-26 (17 months)

To examine the research questions, and minimise bias, the proposed design is a single-blind randomised controlled trial, with two-groups. The aim of this phase will be to respond to research questions such as what are recruitment and retention rates over 6 months; are the trial assessments and interventions acceptable to parents and professionals; are there functional data collection systems enabling future cost effectiveness analysis. This phase will also assess fidelity to the DDP model and whether the care pathways to CAMHS are maintained throughout.

The research team will aim to recruit around 60 families. The potential participants will be identified and approached by their usual service provider. The usual service research administrator will ensure eligible families receive the study participant information leaflet to learn about the study. Once the interest of the family to take part in the trial is confirmed, a research nurse will contact interested families 24 hours later, to discuss the study further and seek consent. Families that confirm their willingness to participate will be invited for two study visits one at baseline, shortly after joining study and second visit after 12 months.

On completion of the baseline data collection, consenting families will be individually randomised 1:1 to DDP or SAU, stratified by site. Individuals who consent to take part will have an equal chance of being randomised to either group. One group will be included in the DDP intervention. The second group will take part in the Services as Usual. The research assistant with responsibility for collecting the data will not know which group participants have been allocated to until the end of the study. The intervention will be delivered by the participant's usual health care team.

Beside the randomised controlled trial, the data will be collected through qualitative research activities to explore social context supporting/hindering child mental health, optimising the contexts of, and processes for, DDP delivery.

Process evaluation

Qualitative work in phase 2 has three main aims:

1. To keep abreast of issues and themes uncovered in Phase 1 in the three feasibility trial sites, to ensure ongoing compliance with guidelines for safe DDP delivery and to explore the social context supporting/hindering child mental health in each site including drivers and barriers to optimal DDP/SAU delivery. 6-10 interviews/focus groups will be conducted with therapists, managers and families across the sites.
2. To explore the same topics from Phase 1 in the seven putative Phase 3 trial sites - optimising the contexts of, and processes for, DDP delivery in those sites and examining compliance with the DDP delivery guidelines established in Phase 1. 18-26 interviews/focus groups will be conducted across the sites.
3. To allow selection of 2-4 additional sites for Phase 3. The number of additional sites required for Phase 3 will be decided based on Phase 2 conversion rates from eligible to consented families and on statistical power considerations based on the standard deviation, in Phase 2, of our principle outcome measure.

Phase 2 will also adopt case study methodology to focus more specifically on the impact of DDP and SAU. The research team will learn through a more in-depth investigation (individual interviews) about participant experience of DDP/SAU and of journeys through service landscapes from the perspectives of the family, therapists, and other key stakeholders involved in the treatment of and care pathways. A small selection of families (2-3 families) will be invited to take part.

Phase 3 Months 27-53 (27 month RCT; (6 month analysis/write-up).

The third phase will continue as a single-blind individually randomised controlled superiority definitive trial. The aim of this phase will be to examine the clinical and cost-effectiveness of DDP for improving child mental health, compared to SAU. The principle outcome will be child's mental health at 12 months post randomisation. The research team will aim to recruit additional 180 families, including phase 2. The study population, interventions, randomisation, data collection, measures, model fidelity and procedures will be as described for Phase 2 unless findings from the process evaluation suggest modifications.

Qualitative evaluation (process evaluation) will continue at the same intensity as Phase 2, with a similar number of interviews/focus groups (24-36 across all sites), to explore delivery drivers/barriers in each service context. The case studies will continue, involving a further 10-12 interviews, to track development over time. The PPCI group and YPAG will have a crucial role in the Process Evaluation, during this phase, in reviewing the qualitative findings with the Process Evaluation Team (PET) and considering how these findings pragmatically feed into future service delivery. Whether or not DDP is eventually found to be cost-effective over services as usual, the process evaluation will yield important information about how mental health services can be safely delivered for maltreated children in different services contexts (i.e. NHS CAMHS, Social Care and Private Practice).

ELIGIBILITY:
Inclusion Criteria:

• Adoptive or permanent foster parents with children aged 5-12 years with symptoms of MAPP or co-occurring mental health conditions and non-psychotherapeutic treatments

Exclusion Criteria:

* Families, otherwise eligible, deemed by therapists as not ready for DDP (usually where therapists have concerns about the ability of carers/parents to create a safe/ nurturing enough environment within which DDP can operate)
* Children currently having another psychotherapy

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Reactive Attachment Disorder and Disinhibited Social Engagement Disorder Assessment (RADA) | 12 months from baseline
  The Reactive Attachment Disorder and Disinhibited Social Engagement Disorder Assessment (RADA) is the only measure of Attachment Disorder symptoms that is well validated against clinician diagnosis in middle childhood. Ii is a diagnostic measure that has algorithms compliant with DSM 5 for Reactive Attachment Disorder (RAD) and Disinhibited Social Engagement Disorder (DSED), and it can also be used as a continuous measure (33-items; scoring range 0-66). Previous research suggests a standard deviation of 10.4 for the RADA. Applying the same assumption as for SDQ (correlation between baseline and follow-up of 0.4, correlation within clusters of 0.03, cluster size of 10, retention rate of 0.72), there will be 90% power to detect a difference in RADA of at least 7.25 with a sample size of 190. Typically developing children usually have very low or zero scores on measures for Attachment Disorders so would consider such a change in RADA to be clinically significant.
Strengths and Difficulties Questionnaire (SDQ) | 12 months from baseline
  Strengths and Difficulties Questionnaire (SDQ) has good sensitivity to change in RCTs. Candidate measures are included for the four problem areas in our logic model: child emotion regulation, parental stress, parent-child relationship functioning and child mental health. The research team estimates that 190 families will be required to determine clinical- and cost effectiveness based on findings from an ongoing trial of maltreated pre-school children, information from clinics using the SDQ to evaluate DDP and SDQ population norms. This aims for 90% power, assumes a clinical difference in SDQ of 4 points, a baseline and 1-year follow-up correlation in SDQ of 0.4, a standard deviation in SDQ of 5.8, an intra-cluster correlation of 0.03 (between families who see the same therapist) and a retention rate of 72%.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Minnis, Professor, Principal Investigator — University of Glasgow
Locations (16):
- United Kingdom (16):
  - Lanarkshire, Lanark, Scotland
  - Vale Valleys and Cardiff Adoption Collaborative, Barry
  - Bedford Borough Council, Bedford
  - Birmingham Children's Trust, Birmingham
  - Bradford District Care Foundation Trust, Bradford
  - One Adoption South Yorkshire, Doncaster
  - Blaenau Gwent County Borough Council, Ebbw Vale
  - South London and Maudsley NHS Foundation Trust, London
  - Norfolk and Suffolk NHS Foundation Trust, Norwich
  - Norfolk County Council, Norwich
  - Nottingham City Council, Nottingham
  - Nottinghamshire County Council (Adoption East Midlands), Nottingham
  - Oxfordshire, Oxford
  - Central Bedfordshire Council, Shefford
  - Hertfordshire County Council, Stevenage
  - Adoption@Heart, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vasileva M, Petermann F. Attachment, Development, and Mental Health in Abused and Neglected Preschool Children in Foster Care: A Meta-Analysis. Trauma Violence Abuse. 2018 Oct;19(4):443-458. doi: 10.1177/1524838016669503. Epub 2016 Sep 22. PMID 27663993
- [Background] Harkess-Murphy E, Macdonald J, Ramsay J. Self-harm and psychosocial characteristics of looked after and looked after and accommodated young people. Psychol Health Med. 2013;18(3):289-99. doi: 10.1080/13548506.2012.712706. Epub 2012 Aug 6. PMID 22867514
- [Background] Font SA, Maguire-Jack K. Pathways from childhood abuse and other adversities to adult health risks: The role of adult socioeconomic conditions. Child Abuse Negl. 2016 Jan;51:390-9. doi: 10.1016/j.chiabu.2015.05.013. Epub 2015 Jun 6. PMID 26059537
- [Background] Duncan AE, Auslander WF, Bucholz KK, Hudson DL, Stein RI, White NH. Relationship between abuse and neglect in childhood and diabetes in adulthood: differential effects by sex, national longitudinal study of adolescent health. Prev Chronic Dis. 2015 May 7;12:E70. doi: 10.5888/pcd12.140434. PMID 25950577
- [Background] Rivenbark JG, Odgers CL, Caspi A, Harrington H, Hogan S, Houts RM, Poulton R, Moffitt TE. The high societal costs of childhood conduct problems: evidence from administrative records up to age 38 in a longitudinal birth cohort. J Child Psychol Psychiatry. 2018 Jun;59(6):703-710. doi: 10.1111/jcpp.12850. Epub 2017 Dec 2. PMID 29197100
- [Background] Burt SA, Hyde LW, Frick PJ, Jaffee SR, Shaw DS, Tremblay R. Commentary: Childhood conduct problems are a public health crisis and require resources: a commentary on Rivenbark et al. (). J Child Psychol Psychiatry. 2018 Jun;59(6):711-713. doi: 10.1111/jcpp.12930. PMID 29808490
- [Background] Denham SA, Bassett HH, Sirotkin YS, Brown C, Morris CS. "No-o-o-o Peeking": Preschoolers' Executive Control, Social Competence, and Classroom Adjustment. J Res Child Educ. 2015 Apr 1;29(2):212-225. doi: 10.1080/02568543.2015.1008659. PMID 26166925
- [Background] Li D, Chng GS, Chu CM. Comparing Long-Term Placement Outcomes of Residential and Family Foster Care: A Meta-Analysis. Trauma Violence Abuse. 2019 Dec;20(5):653-664. doi: 10.1177/1524838017726427. Epub 2017 Aug 31. PMID 29333987
- [Background] Luchenski S, Maguire N, Aldridge RW, Hayward A, Story A, Perri P, Withers J, Clint S, Fitzpatrick S, Hewett N. What works in inclusion health: overview of effective interventions for marginalised and excluded populations. Lancet. 2018 Jan 20;391(10117):266-280. doi: 10.1016/S0140-6736(17)31959-1. Epub 2017 Nov 12. PMID 29137868
- [Background] Dozier M, Peloso E, Lewis E, Laurenceau JP, Levine S. Effects of an attachment-based intervention on the cortisol production of infants and toddlers in foster care. Dev Psychopathol. 2008 Summer;20(3):845-59. doi: 10.1017/S0954579408000400. PMID 18606034
- [Background] Nelson CA, Fox NA, Zeanah CH. Developmental Psychopathology 2016:1-37.
- [Background] Wright B, Barry M, Hughes E, Trepel D, Ali S, Allgar V, Cottrill L, Duffy S, Fell J, Glanville J, Glaser D, Hackney L, Manea L, McMillan D, Palmer S, Prior V, Whitton C, Perry A, Gilbody S. Clinical effectiveness and cost-effectiveness of parenting interventions for children with severe attachment problems: a systematic review and meta-analysis. Health Technol Assess. 2015 Jul;19(52):vii-xxviii, 1-347. doi: 10.3310/hta19520. PMID 26177494
- [Background] National Collaborating Centre for Mental Health (UK). Children's Attachment: Attachment in Children and Young People Who Are Adopted from Care, in Care or at High Risk of Going into Care. London: National Institute for Health and Care Excellence (NICE); 2015 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK338143/ PMID 26741018
- [Background] Looked-after children and young people. London: National Institute for Health and Care Excellence (NICE); 2021 Oct 20. Available from http://www.ncbi.nlm.nih.gov/books/NBK575858/ PMID 34941234
- [Background] Dinkler L, Lundstrom S, Gajwani R, Lichtenstein P, Gillberg C, Minnis H. Maltreatment-associated neurodevelopmental disorders: a co-twin control analysis. J Child Psychol Psychiatry. 2017 Jun;58(6):691-701. doi: 10.1111/jcpp.12682. Epub 2017 Jan 17. PMID 28094432
- [Background] Cecil CA, Viding E, Fearon P, Glaser D, McCrory EJ. Disentangling the mental health impact of childhood abuse and neglect. Child Abuse Negl. 2017 Jan;63:106-119. doi: 10.1016/j.chiabu.2016.11.024. Epub 2016 Nov 30. PMID 27914236
- [Background] . Van der Kolk BA. Psychiatric annals 2017;35:401-8.
- [Background] Kay C, Green J. Reactive attachment disorder following early maltreatment: systematic evidence beyond the institution. J Abnorm Child Psychol. 2013 May;41(4):571-81. doi: 10.1007/s10802-012-9705-9. PMID 23250477
- [Background] Minnis H. Maltreatment-associated psychiatric problems: an example of environmentally triggered ESSENCE? ScientificWorldJournal. 2013 Apr 17;2013:148468. doi: 10.1155/2013/148468. Print 2013. PMID 23710133